CLINICAL TRIAL: NCT05986006
Title: Fusion Status of Machined Allograft Versus Iliac Crest Allograft in Anterior Cervical Discectomy and Fusion: A Randomized Controlled Trial
Brief Title: Fusion Status After ACDF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHIL22D.618
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Spine Fusion; Spine Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Cervical Discectomy and Fusion (ACDF) w/Machined Allograft (Active Comparator): Participant will undergo primary, elective one-level to four-level ACDF and will be randomized to machined bone allograft
  Interventions: Procedure: Anterior Cervical Disc Fusion (ACDF) Surgery w/ machined bone allograft
- Anterior Cervical Discectomy and Fusion (ACDF) w/Iliac Crest Allograft (Active Comparator): Participant will undergo primary, elective one-level to four-level ACDF and will be randomized to iliac crest bone allograft
  Interventions: Procedure: Anterior Cervical Disc Fusion (ACDF) Surgery w/ Iliac Crest Bone Graft

INTERVENTIONS:
Procedure: Anterior Cervical Disc Fusion (ACDF) Surgery w/ machined bone allograft — Participant will undergo primary, elective one-level to four-level ACDF using machined bone allograft
  Arms: Anterior Cervical Discectomy and Fusion (ACDF) w/Machined Allograft
Procedure: Anterior Cervical Disc Fusion (ACDF) Surgery w/ Iliac Crest Bone Graft — Participant will undergo primary, elective one-level to four-level ACDF using iliac crest bone allograft
  Arms: Anterior Cervical Discectomy and Fusion (ACDF) w/Iliac Crest Allograft

SUMMARY:
Pseudarthrosis, a failure of bony fusion, is one of the most common causes of revision surgery following anterior cervical discectomy and fusion (ACDF). The interbody spacer is an important component of bony fusion in ACDF, and we aim to compare machined allograft spacers versus iliac crest allograft in a randomized controlled trial.

DETAILED DESCRIPTION:
Pseudarthrosis, a failure of bony fusion, is one of the most common causes of revision surgery following anterior cervical discectomy and fusion (ACDF). The interbody spacer is an important component of bony fusion in ACDF, and we aim to compare machined allograft spacers versus iliac crest allograft in a randomized controlled trial. We hypothesize that iliac crest allograft will improve anterior cervical discectomy and fusion arthrodesis rates and diminish the amount of intervertebral graft resorption when compared to off-the-shelf machined allografts

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older
* preoperative diagnosis of cervical radiculopathy and/or cervical myelopathy.

Exclusion Criteria:

* patients undergoing a revision cervical procedure
* current smokers
* patient with surgical indications of tumor, infection, or trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-08-07 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Improved participant reported outcome measures (PROMs)-1 | 2 years
  Investigators will ask participants to complete the Short Form-12 survey (SF-12) at 3 months, 6 months, 12 months, and 24 months following surgery
Improved participant reported outcome measures (PROMs)-2 | 2 years
  Investigators will ask participants to complete the Visual Analog Score (VAS) for Neck and Arm, Neck Disability Index (NDI), at 3 months, 6 months, 12 months, and 24 months following surgery
Improved participant reported outcome measures (PROMs)-3 | 2 years
  Investigators will ask participants to complete the modified Japanese Orthopaedic Association (mJOA) score) at 3 months, 6 months, 12 months, and 24 months following surgery
Fusion status after surgery | 2 years
  Fusion status will be assessed using Postoperative x-rays (AP, lateral, flexion, extension) which will be taken at 3 months, 6 months, 12 months, and 24 months following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States